CLINICAL TRIAL: NCT07160218
Title: The Effect of Trans-cranial Direct Current Stimulation and Cognitive Rehabilitation on Cognitive Functions and Neuronal Plasticity inPatients With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Effects of tDCS and Cognitive Rehabilitation on Cognition and Neural Plasticity in MS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehrdad Roozbeh, Assistant Professor of Neurology, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.SBMU.PHNS.REC.1402.121
Record Dates: First submitted 2025-08-26; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS (Experimental): A 30-minute tDCS session with the cathode placed over the left dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: tDCS
- tDCS+Cognitive training (Experimental): A 30-minute tDCS session with the cathode over the left DLPFC combined with computer-based cognitive rehabilitation training
  Interventions: Device: tDCS; Device: Cognitive Rehabilitation
- Sham tDCS (Sham Comparator): Sham stimulation applied over the left DLPFC, mimicking the sensation of tDCS without delivering active current
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: tDCS — A 30-minute tDCS session with the cathode placed over the left dorsolateral prefrontal cortex (DLPFC), delivered in 10 sessions over 2 weeks. This protocol targets cognitive improvement in MS patients
  Arms: tDCS; tDCS+Cognitive training
Device: Cognitive Rehabilitation — computer-based cognitive rehabilitation exercises. Conducted in 10 sessions over 2 weeks to enhance attention, memory, and neuroplasticity in MS patients.
  Arms: tDCS+Cognitive training
Device: Sham tDCS — Sham stimulation applied over the left DLPFC for 30 minutes, mimicking the sensation of tDCS without delivering active current, over 10 sessions, used as control to blind participants to the intervention
  Arms: Sham tDCS

SUMMARY:
The goal of this clinical trial is to evaluate whether transcranial direct current stimulation (tDCS) and cognitive rehabilitation can improve cognitive functions and neuronal plasticity in patients with multiple sclerosis (MS). The participant population consists of MS patients (both sexes, adults), who commonly experience cognitive impairment in addition to physical and psychological symptoms.

The main questions it aims to answer are:

Does tDCS applied over the left dorsolateral prefrontal cortex improve cognitive abilities in MS patients?

Does the combination of tDCS and cognitive rehabilitation enhance neuroplasticity, as measured by DTI, BDNF levels, and acetylcholinesterase activity?

ELIGIBILITY:
Inclusion Criteria:

Age between 20 and 50 years.

Diagnosed with relapsing-remitting multiple sclerosis (RRMS).

Mild disability, defined as EDSS < 5.

Patients who attended the neurology clinic and are willing to participate.

Exclusion Criteria:

Presence of psychiatric disorders requiring treatment with neuroleptics.

History of seizures.

Left-handed individuals.

Recent MS relapse requiring steroid treatment.

Pregnant women.

History of brain surgery or presence of intracranial clips.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in verbal memory performance measured by California Verbal Learning Test-II (CVLT-II) | Baseline and immediately after 10 intervention sessions
  The CVLT-II assesses verbal learning and memory through a word recall task. Scores include total recall, short-delay recall, and long-delay recall. Assessments will be conducted at baseline and after 4 weeks of intervention.
Change in attention performance measured by Integrated Visual and Auditory Continuous Performance Test (IVA-2) | Baseline and immediately after 10 intervention sessions
  The IVA-2 evaluates visual and auditory attention and response control. Scores include full-scale attention quotient, visual attention, auditory attention, and response control. Assessments will be conducted at baseline and post-intervention to assess changes in attention performance
Change in visuospatial memory performance measured by Rey-Osterrieth Complex Figure Test | Baseline and immediately after 10 intervention sessions
  The Rey-Osterrieth Complex Figure Test evaluates visuospatial constructional ability and memory. Participants copy a complex figure (copy trial) and then reproduce it from memory immediately and after a delay. Assessments will be conducted at baseline and after completion of the tDCS intervention to assess changes in visuospatial memory performance.
Change in serum BDNF levels (ng/mL) | Baseline and immediately after 10 intervention sessions
  Serum brain-derived neurotrophic factor (BDNF) concentration will be measured using an enzyme-linked immunosorbent assay (ELISA). Blood samples will be collected at baseline and after completion of the tDCS intervention. Changes in BDNF levels will be analyzed to assess neuroplasticity.
Change in white matter integrity measured by Diffusion Tensor Imaging (DTI) | Baseline and immediately after 10 intervention sessions
  White matter integrity will be assessed using DTI MRI scans. Primary metrics include Fractional Anisotropy (FA) and Mean Diffusivity (MD) in predefined brain regions. Scans will be performed at baseline and after completion of the tDCS intervention to evaluate neuroplasticity-related changes
Change in acetylcholinesterase (AChE) activity in blood (U/mL) | Baseline and immediately after 10 intervention sessions
  Acetylcholinesterase activity will be measured in blood samples using a spectrophotometric enzymatic assay. Samples will be collected at baseline and after completion of the tDCS intervention. Changes in AChE activity will be analyzed to assess cholinergic system function and neuroplasticity.

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Beheshti University of Medical Science, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available to qualified researchers. Data sharing will occur after the publication of the primary study results. Requests for data access will be considered on a case-by-case basis and can be initiated by contacting the corresponding author. Data will be shared under a data use agreement to ensure appropriate use and confidentiality